CLINICAL TRIAL: NCT00783042
Title: A Randomised, Double-Blind, Placebo-Controlled Study to Evaluate the Transthoracic Doppler Echocardiography Method as a Non-Invasive Method for Coronary Function Measurements; Ability to Detect Short-Term Statin Effects in Patients With Increased Cardiovascular Risk
Brief Title: Exploratory Study of Coronary Flow Reserve Measurements, a Non-Invasive Method for Coronary Function Measurements
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Björn Carlsson MD, PhD, Medical Science Director, Clinical Discovery Team CV/GI, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D1840M00006
Record Dates: First submitted 2008-10-30; First posted 2008-10-31 (Estimated); Last update posted 2009-06-30 (Estimated); Status verified 2009-06

CONDITIONS: Atherosclerosis; Inflammatory Activity in Coronary Arteries
Keywords: TTDE-CFR; coronary artery function; cardiovascular biomarkers; rosuvastatin; Crestor
MeSH Terms: conditions — Atherosclerosis | interventions — Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator)
  Interventions: Drug: Rosuvastatin
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Rosuvastatin — 40 mg, tablet, oral, once daily for 1 (double blind) +2 months (open).
  Other Names: Crestor
  Arms: 1
Drug: Placebo — Tablet, oral, once daily for 1 month (double blind)
  Arms: 2

SUMMARY:
The aim of this study is to investigate whether the non-invasive ultrasound method for assessment of coronary blood flow, transthoracic Doppler echocardiography-coronary flow reserve (TTDE-CFR), can be used to measure drug effects.

ELIGIBILITY:
Inclusion Criteria:

* Males aged 45-75 years or females aged 60-75 years inclusive
* Carotid and/or femoral atherosclerotic plaque, as assessed by carotid ultrasound examination within the last 5 years
* Abnormal concentrations of lipids or lipoproteins in the blood
* Provision of signed informed consent

Exclusion Criteria:

* Treatment with statins or other lipid-lowering drugs, e.g. fibrates, nicotinic acid, cholesterol absorption inhibitor, within the last 6 months before randomisation
* Current smoking or snuff tobacco use
* Major CV event (myocardial infarction (MI), stroke/ transitory ischemic attack (TIA), Acute Coronary Syndrome (ACS), revascularisation) within the last 6 months before randomisation
* Symptomatic carotid stenosis, atrioventricular (AV) block, QT-prolongation, atrial fibrillation, sinus node disease (such as sick sinus syndrome or symptomatic bradycardia), chronic obstructive pulmonary disease (COPD) or asthma

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2008-10; Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Change in CFR peak velocity within rosuvastatin group after 1 month of treatment compared to baseline | Baseline and after 1 month of treatment
Comparison of treatment effects on CFR peak velocities between groups after 1 month of treatment | Baseline and after 1 month of treatment

SECONDARY OUTCOMES:
Changes in CFR peak velocity within the rosuvastatin group after 3 months compared to baseline and to 1 month | Bseline, after 1 month and after 3 months of treatment
Changes in other CFR parameters after one month rosuvastatin or placebo treatment; comparisons within groups and between groups | Baseline and after 1 month of treatment
Changes in plasma lipids, lipoproteins and other cardiovascular biomarkers after 1 month of treatment with rosuvastatin or placebo; comparisons within groups and between groups | Baseline and after 1 month of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Björn Fagerberg, MD, Professor, Principal Investigator — Wallenberg LaboratorySahlgrenska University Hospital, S-413 45 Göteborg; Maria Leonsson-Zachrissson, MD, Study Chair — AstraZeneca R&D Mölndal
Locations (1):
- Research Site, Gothenburg, Sweden